CLINICAL TRIAL: NCT07100639
Title: From Exposome to Health Outcomes: A Population-Based Approach to Understanding and Mitigating Early Menopause in Singapore's Diverse Communities
Brief Title: Singapore Population Research on Integrated exposoMe & Early Menopause
Acronym: SG-PRIME
Status: Not yet recruiting | Type: Observational
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Kothandaraman Narasimhan, Ph.D., Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Other Study IDs: 2050-50; MOH-001786-00 (Other: NMRC, Singapore)
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Early Menopause
Keywords: early menopause; environment; pollution; exposome
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SG-PRIME: no interventions

SUMMARY:
Brief Summary

The goal of this observational study is to learn how environmental factors, lifestyle choices, and social conditions affect the timing of menopause in Asian women aged 40-50 years living in Singapore. The main aims of the project are the following:

* Do environmental pollutants and lifestyle exposures contribute to earlier menopause in Asian women?
* What biological changes occur when women are exposed to harmful environmental factors during menopause transition?

Participants will be followed for 18 months and will complete questionnaires about their health history, lifestyle, diet, and environmental exposures. Participants will provide blood, urine, stool, hair, and nail samples for laboratory analysis and undergo basic health assessments including weight, blood pressure, and bone density measurements. Participants will wear activity monitors and air pollution sensors for 7 days and attend follow-up visits at 6 months, 12 months, and 18 months to track changes in their health. This data will be obtained during the baseline visit.

DETAILED DESCRIPTION:
Detailed Description

Background and Rationale: Early menopause, defined as cessation of ovarian function before age 45, affects approximately 5-12% of women globally and is associated with increased risks of cardiovascular disease, osteoporosis, and cognitive decline. Growing evidence suggests that environmental exposures, including persistent organic pollutants, air pollution, and endocrine-disrupting chemicals, may accelerate ovarian aging and contribute to earlier menopausal timing. The exposome concept involves the totality of environmental exposures experienced by individuals throughout their lifetimes, including chemical, physical, biological, and social factors.

Study Hypothesis We hypothesize that combined exposure to environmental pollutants, lifestyle factors, and social conditions accelerates biological aging processes and leads to earlier menopause onset in women. These exposome effects are mediated through changes in gene expression patterns, metabolic profiles, and gut microbiome composition, ultimately increasing the risk of adverse health outcomes.

Study Design: This is a prospective observational cohort study employing a longitudinal design with 18-month follow-up. The study integrates comprehensive exposome assessment with multi-omics profiling to investigate the complex relationships between environmental factors and menopausal health outcomes in a multi-ethnic Asian population.

Population and Setting: Four hundred women aged 40-50 years will be recruited from diverse communities across Singapore. Participants must have experienced no menstruation for the last 2 months or irregular menstrual cycles in the last 6 months, be proficient in English, and plan to reside in Singapore for the study duration. The study will include Chinese, Malay, and Indian ethnicities reflecting Singapore's demographic composition.

Data Collection Methods: Exposome characterization includes external environmental monitoring through air pollution assessment, climate data collection, green space quantification, and personal exposure measurement using wearable devices. Biological samples including blood, urine, stool, hair, and nail specimens will undergo multi-omics analysis encompassing metabolomics, lipidomics, epigenetics, transcriptomics, and microbiome profiling. Clinical assessments include anthropometric measurements, blood pressure monitoring, and bone density evaluation.

Analysis Plan: Multi-layered analytical approaches will include exposome-wide association studies, machine learning techniques for predictive modeling, and causal inference methods to examine relationships between exposome factors and menopausal outcomes. Advanced statistical methods will account for the high-dimensional nature of exposome data and temporal relationships between exposures and health outcomes.

Eligibility Criteria

Inclusion Criteria:

* Female participants aged 40-50 years
* No menstruation for the last 2 months or irregular menstrual cycles in the last 6 months
* Chinese, Malay, or Indian ethnicity
* Proficient in English language
* Planning to reside in Singapore for next 2 years
* Willing to provide informed consent and comply with study procedures

Exclusion Criteria:

* In menopause (12 consecutive months without menstruation)
* Currently pregnant or planning to conceive
* History of bilateral oophorectomy and/or hysterectomy
* Currently receiving hormone therapy, including estradiol replacement therapy or oral contraceptives
* Diagnosed with premature ovarian insufficiency before 40 years of age
* Diagnosis of autoimmune conditions and/or chromosomal abnormalities known to affect ovarian function
* Diagnosis of severe cognitive impairment and/or mental disorders
* Received cancer treatment in the past 12 months

Target Sample Size 400 participants

ELIGIBILITY:
Inclusion Criteria:

Female participants aged 40-50 years No menstruation for the last 2 months or irregular menstrual cycles in the last 6 months Chinese, Malay, or Indian ethnicity Proficient in English language Planning to reside in Singapore for next 2 years Willing to provide informed consent and comply with study procedures

Exclusion Criteria:

In menopause (12 consecutive months without menstruation) Currently pregnant or planning to conceive History of bilateral oophorectomy and/or hysterectomy Currently receiving hormone therapy, including estradiol replacement therapy or oral contraceptives Diagnosed with premature ovarian insufficiency before 40 years of age Diagnosis of autoimmune conditions and/or chromosomal abnormalities known to affect ovarian function Diagnosis of severe cognitive impairment and/or mental disorders Received cancer treatment in the past 12 months

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women experiencing perimenopausal transition characterized by irregular menstrual patterns and hormonal fluctuations, stratified by age groups (40-45 years and 46-50 years) and ethnicity to ensure representative sampling of Singapore's multi-ethnic population.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-06 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Early menopause | 18 months
Time to menopause onset | 18 months
  • Menopausal symptom severity score using standardized assessment tools

IPD SHARING:
Plan to Share IPD: Undecided